CLINICAL TRIAL: NCT01730612
Title: Pilot Study for Optimization of Immuno-PET Pretargeted With Anti-CEA Bispecific Antibody X Anti-HSG TF2 and the Peptide IMP-288 Radiolabeled With Gallium-68 -Pharmacokinetic and Imaging for Patients With a Recurrence of HER2 Negative Breast Carcinoma Expressing CEA
Brief Title: ImmunoTEP au 68-Ga- IMP-288 for Patients With a Recurrence of HER2 Negative Breast Carcinoma Expressing CEA
Acronym: iTEPsein
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD/10/04-O
Record Dates: First submitted 2012-11-12; First posted 2012-11-21 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2017-05

CONDITIONS: HER2 Negative Breast Carcinoma Expressing CEA
Keywords: ImmunoTEP; HER2 negative; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: TF2 - 68 Ga-IMP-288: — ImmunoTEP
  Other Names: TF2: trivalent recombinant humanized antibody recognizing the ACE and the peptide histamine-succinyl-glycine IMP-288 (HSG); 68 Ga-IMP-288: di-HSG peptide-DOTA-labeled with Gallium 68

SUMMARY:
Main objective: To determine the optimal molar doses of the biospecific antibody TF2 and 68 Ga-IMP-288 and the optimal time for pretargeting for immuno-PET in patients with breast carcinoma.

Secondary objectives: To study the sensitivity of the immuno-PET, compare its performance to standard imaging methods, evaluate the safety of 150 MBq of 68 Ga-IMP-288; study the development of immunization against TF2 or complex TF2-IMP-288;

DETAILED DESCRIPTION:
* 4 or 5 cohorts of 3 patients receiving different doses of TF2 IMP-288 with different interval time. A last cohort (4 or 5 ): maximum of 21 additional patients with the optimal schedule.

Cohort I: TF2 120 nmol / 6 nmol IMP-288 / 24 hours

Cohort II: based on the results of the cohort I :

1. Good signal of the tumor but high background: increased interval time, 120 nmol TF2 / 6 nmol of IMP-288 / 30 hours
2. Low signal of the tumor: reduction of the interval time, 120 nmol TF2 / 6 nmol IMP-288 / 18 hours
3. Good signal of the tumor and good background signal : dose reduction, 60 nmol TF2 / 3nmol IMP- 288 / 24 hours

   Cohort III: based on results of cohort II:

   - Good signal of the tumor : dose reduction, 120 nmol TF2 / 3 nmol IMP-288 / 30 h

   Cohort IV : based on results of cohort III Cohort V : Based on results of cohort IV

   • A last Cohort (VI) : 19 patients with the optimal schedule of injection : 120 nmol TF2 / 3 nmol IMP-288 / 30 h or 120 nmol TF2 / 6 nmol IMP-288 / 30 h

   • In the four weeks prior to the immuno-PET:

   - Clinical examination,

   - CEA and CA15-3,

   - thoraco abdominal pelvic scan, bone scan, FDG-PET,

   - immunohistochemistry ACE on the tumor if possible,

   - Anti-Antibodies if the patient has already received MAb,

   - pregnancy test within 2 days prior to immuno-PET,

   - (creatinine > 2.5 normal) D0: Injection of TF2 D1 to D4: injection of 68 Ga-IMP-288 (depending of the cohort) D0 to D4 : pharmacokinetics, imaging

   Evaluation at 1 month of Immuno-PET:

   • Assessment of the clinical oncologist and

   - histological biopsy and / or surgery performed according to the results of imaging and assessment of the potential clinical impact

   Evaluation at 3 and 6 months of immuno-PET:

   based on the results of immuno-PET, evaluation and therapeutic decision of the oncologist,

   - Imaging (ultrasound, bone scintigraphy, CT or PET FDG),

   - markers
   * Anti-Antibody Search
   * For patient with a cancer treatment a new immuno-PET can be proposed

ELIGIBILITY:
Inclusion Criteria:

* Breast carcinoma, HER2 + (Dako) and HER2 + (fish) metastatic at least after treatment with current consensus
* ≥ 18 years
* Negative pregnancy test for women of childbearing age. Women of childbearing age should take effective contraception continuously for 3 months.
* Karnofsky ≥ 70 or ECOG 0-1

  •• ACE of the tumor by immunohistochemistry or positive plasma CEA ≥ 10 ng / mL
* At least one measurable lesion on CT
* creatinine < 2.5
* Informed consent signed
* Social insurance

Exclusion Criteria:

* Pregnancy or breastfeeding

  * Serious illness or co-morbidity risk assessed
  * History of cancer within 5 years except skin cancer other than melanoma or carcinoma in situ of the cervix
  * Presence of anti-antibodies in patients who have previously received antibodies
  * Known hypersensitivity to antibodies or proteins
  * intellectual disability to sign the informed consent
  * Not controlled diabetes
  * Persons protected by law

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
evaluation of the tumor targeting (no Unit) and signal / noise ratio (no unit) by the immunoTEP with TF2 and 68-Ga-IMP-288 | One week
  Pk blood after injections of TF2 and 68 Ga-IMP-288 and PET imaging semi-quantification with 60 to 120 minutes after injection of 68 Ga-IMP-288

SECONDARY OUTCOMES:
Sensibility, tolerance | 6 months after immunoTEP
  sensitivity of the immuno-PET and compare its performance to standard imaging methods, pathological data if available data or imaging follow-up of at least 6 months by RECIST and EORTC
To study the contribution of immnoTEP to assess early response to treatment, compare its performance to standard imaging methods | month 6
  6 weeks after initiation of treatment of metastases (after the first iTEP), a second _iTEP with a therapeutic evaluation will be carried out. The examination requirements are identical to those of the first immunoTEP.
  this second iITEP will be evaluated in regard of imaging assessment performed routinely (TAP scanner, FDG-PET, CA15-3 and CEA)

OTHER OUTCOMES:
• To assess the tolerance of 150 MBq of 68 Ga-IMP-288 | 6 months
To search for the development of immunization with TF2 and the complex TF2-IMP-288: ELISA | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: francoise Bodere, PhD, MD, Principal Investigator — Nantes Hospital
Locations (2):
- France (2):
  - Hospital, Nantes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain